CLINICAL TRIAL: NCT05749367
Title: Lateral Femoral Cutaneous Nerve and Pericapsular Nerve Group (PENG) Blocks Versus Suprainguinal Fascia Iliaca Block in Postoperative Analgesia of Hip Fractures: a Prospective, Controlled, Randomized and Double Blind Study
Brief Title: Lateral Cutaneous Nerve and PENG Blocks Versus Suprainguinal Fascia Iliaca Block in Post-op Analgesia of Hip Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, Professor of Surgery Department at Medical School of Universidade Federal de Minas Gerais. Ph.D, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE:42438721.1.0000.5129
Record Dates: First submitted 2023-02-08; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia, Conduction
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized and double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the control group, patients will undergo SIFIB with ropivacaine and to maintain the masking they will also undergo PENG and LFCNB with saline solution (sham block). In the experimental group, patients will receive ropivacaine in the PENG block associated with LFCNB and saline solution in the SIFIB. All the work of randomization, editing of the spreadsheet, manipulation of the envelopes, as well as the confidential tabulation of the data during collection will be done by an assistant who will not participate in the anesthesia or data collection. The opening of the envelopes and the preparation of the material for anesthesia will also be done by an assistant who will not participate in the evaluation of the outcomes. The researcher will perform all the procedures and data collection and will not know which group the participant belongs to. The patient will also not know in which group he or she is allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprainguinal Fascia Iliaca Block Group (Active Comparator): Patients will undergo SIFIB with ropivacaine and PENG plus LFCNB with saline solution.
  Interventions: Drug: Ropivacaine + saline solution
- PENG Block + Lateral Femoral Cutaneous Nerve Block Group (Experimental): Patients will undergo SIFIB with saline solution and PENG plus LFCNB ropivacaine.
  Interventions: Drug: Saline solution + Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine + saline solution — SIFIB with 30 ml of 0.5% ropivacaine and PENG Block plus LFCNB with 20 ml and 10 ml of saline solution, respectively.
  Other Names: Naropin + saline solution
  Arms: Suprainguinal Fascia Iliaca Block Group
Drug: Saline solution + Ropivacaine — SIFIB with 30 ml of saline solution and PENG Block plus LFCNB with 20 ml and 10 ml of 0,5% ropivacaine, respectively.
  Other Names: Saline solution + Naropin
  Arms: PENG Block + Lateral Femoral Cutaneous Nerve Block Group

SUMMARY:
Postoperative pain in hip fractures is challenging and requires adequate management. Peripheral nerve blocks are already known as superior than systemic analgesia in this scenario, but the best analgesic regional technique is still unknown. The investigators propose a study to compare the postoperative analgesia of hip fractures between pericapsular nerve group block plus lateral femoral cutaneous nerve block and suprainguinal fascia iliaca block

DETAILED DESCRIPTION:
Postoperative pain in hip fractures is challenging and requires adequate management. In this scenario, peripheral nerve blocks present superior results to systemic analgesia, minimizing the use of opioids and their adverse effects. The lumbar plexus is responsible for the nociception of the hip joint through the femoral, obturator, and accessory obturator nerves, besides being responsible for the sensory innervation of the lateral aspect of the thigh through the lateral femoral cutaneous nerve. Due to this intricate network, several regional techniques have already been proposed. However, the best analgesic approach is still unknown. Ultrasound-guided suprainguinal fascia iliaca block (SIFIB), which addresses the femoral and lateral femoral cutaneous nerves, and ultrasound-guided pericapsular nerve group block (PENG), which addresses terminal branches of the femoral and accessory obturator nerves, are techniques currently used successfully in the context of analgesia for hip surgery. PENG block generates less motor impairment of the quadriceps, which can be significant in terms of mobility and rehabilitation. Both techniques show similar analgesic results in the still scarce literature, but SIFIB has shown slight advantage in some scenarios. However, the PENG block does not reach the lateral cutaneous nerve, which may lead to greater postoperative pain perception. In an attempt to fill this knowledge gap, the investigators propose a study to analyze whether the association between PENG block and lateral femoral cutaneous nerve block (LFCNB) promotes postoperative analgesia equal to SIFIB in a population of adults with hip fractures. This will be a prospective, controlled, randomized, double blind study. Patients with hip fractures (femoral neck, transtrochanteric and subtrochanteric) who will undergo surgical treatment (hip arthroplasty and osteosynthesis with intramedullary nails or screws) will be recruited and randomly allocated into two groups: control (C) and experimental (E). In group C, patients will undergo SIFIB with 30 ml of 0.5% ropivacaine, and to maintain blinding they will also undergo PENG and LFCNB with 20 ml and 10 ml of saline, respectively. In group E, patients will receive the PENG block associated with LFCNB, with 20ml + 10ml of 0.5% ropivacaine, respectively, and 30 ml of saline solution in the SIFIB. After performing the blocks, all patients will undergo spinal anesthesia, with intrathecal injection of 10mg of 0.5% isobaric bupivacaine. As a primary objective, the investigators will evaluate dynamic pain (passive elevation of the leg at 15°) using the Numeric Rating Scale (0-10), 6 hours, 12 hours and 24 hours after spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip fractures who will undergo surgical treatment.
* Adults over 18 years.
* American Society of Anesthesiology physical status 1 to 3.
* Body mass index (BMI) < 35 Kg/m2.

Exclusion Criteria:

* Local anesthetic allergy
* Coagulopathy
* American Society of Anesthesiology physical status ≥ 4,
* Dementia
* Peripheral polyneuropathy
* Pregnancy
* Chronic opioid use (> 3 months)
* BMI >35 Kg/m2
* Stroke with lower limb motor sequelae
* Patient refusal/withdrawal
* Those whose spinal anesthesia has been changed to general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03-06 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Dynamic Post-op Hip Pain | 6 hours after spinal anesthesia.
  To assess dynamic hip pain (passive leg elevation at 15°) in postoperative period using the Numeric Rating Scale (0-10), on which patients rate their current pain intensity from (no pain) to 10 (worst possible pain).
Dynamic Post-op Hip Pain | 12 hours after spinal anesthesia
  To assess dynamic hip pain (passive leg elevation at 15°) in postoperative period using the Numeric Rating Scale (0-10), on which patients rate their current pain intensity from (no pain) to 10 (worst possible pain).
Dynamic Post-op Hip Pain | 24 hours after spinal anesthesia
  To assess dynamic hip pain (passive leg elevation at 15°) in postoperative period using the Numeric Rating Scale (0-10), on which patients rate their current pain intensity from (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Post-op Hip Pain at Rest | 6 hours, 12 hours and 24 hours after spinal anesthesia.
  To evaluate hip pain at rest in postoperative period using the Numeric Rating Scale (0-10), on which patients rate their current pain intensity from ) (no pain) to 10 (worst possible pain)..
Quadriceps muscle strength measured by dynamometry in newton (N). | 6 hours, 12 hours and 24 hours after spinal anesthesia.
  To test the quadriceps muscle strength by dynamometry (Med Force hand-held push dynamometer, tHHD, MED.DOR Ltd., Governador Valadares, Brazil) in newton.
Quadriceps muscle strength index | 6 hours, 12 hours and 24 hours after spinal anesthesia.
  To calculate quadriceps muscle strength index by the ratio between the strengths (collected by dynamometry) of the non-operated and operated lower limbs.
Total intravenous morphine dose in milligram over 24 hours | 24 hours
  To quantify the total rescue morphine dose (or morphine equivalent) in mg over 24h.
Time of the first morphine order in minutes | 24 hours
  To record the time of the first morphine order in minutes after the spinal anesthesia
Incidence of opioid side effects | 24 hours
  To record the incidence of opioid side effects - nausea/vomiting, pruritus, urinary retention and respiratory depression
Incidence of blockades complications | 24 hours
  To record the incidence of blockades complications - vascular puncture, hematoma, local anesthetic toxicity and nerve injury.
Incidence of delirium | 24 hours
  To evaluate altered cognition and conclude as positive or negative.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo SG Oliveira, MD, Principal Investigator — Hospital Municipal Odilon Behrens - Belo Horizonte/Brazil and Universidade Federal de Minas Gerais
Locations (1):
- Hospital Odilon Behrens, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043
- [Background] Bugada D, Bellini V, Lorini LF, Mariano ER. Update on Selective Regional Analgesia for Hip Surgery Patients. Anesthesiol Clin. 2018 Sep;36(3):403-415. doi: 10.1016/j.anclin.2018.04.001. Epub 2018 Jul 11. PMID 30092937
- [Background] Vermeylen K, Desmet M, Leunen I, Soetens F, Neyrinck A, Carens D, Caerts B, Seynaeve P, Hadzic A, Van de Velde M. Supra-inguinal injection for fascia iliaca compartment block results in more consistent spread towards the lumbar plexus than an infra-inguinal injection: a volunteer study. Reg Anesth Pain Med. 2019 Feb 22:rapm-2018-100092. doi: 10.1136/rapm-2018-100092. Online ahead of print. PMID 30798268
- [Background] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Background] Morrison C, Brown B, Lin DY, Jaarsma R, Kroon H. Analgesia and anesthesia using the pericapsular nerve group block in hip surgery and hip fracture: a scoping review. Reg Anesth Pain Med. 2021 Feb;46(2):169-175. doi: 10.1136/rapm-2020-101826. Epub 2020 Oct 27. PMID 33109730
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085
- [Background] Lin DY, Morrison C, Brown B, Saies AA, Pawar R, Vermeulen M, Anderson SR, Lee TS, Doornberg J, Kroon HM, Jaarsma RL. Pericapsular nerve group (PENG) block provides improved short-term analgesia compared with the femoral nerve block in hip fracture surgery: a single-center double-blinded randomized comparative trial. Reg Anesth Pain Med. 2021 May;46(5):398-403. doi: 10.1136/rapm-2020-102315. Epub 2021 Feb 26. PMID 33637625
- [Background] Macedo MC, Souza MA, Ferreira KR, Campos LO, Souza ISO, Barbosa MA, Brito CJ, Intelangelo L, Barbosa AC. Validity and Test-Retest Reliability of a Novel Push Low-Cost Hand-Held Dynamometer for Knee Strength Assessment during Different Force Ranges. Diagnostics (Basel). 2022 Jan 13;12(1):186. doi: 10.3390/diagnostics12010186. PMID 35054353